CLINICAL TRIAL: NCT03982823
Title: Comparison of Stapled and Hand-Sewn Sleeve Gastrectomy, Retrospective Study
Brief Title: Comparison of Stapled and Hand-Sewn Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Serdar Kırmızı, M.D., Fellow at the Department of Gastroenterology Surgery, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/33
Record Dates: First submitted 2019-05-23; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; surgical stapling; suture techniques; natural orifice surgery; transoral; mini-laparoscopy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Stapled Sleeve Gastrectomy Group and Hand-Sewn Sleeve Gastrectomy Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hand-Sewn Sleeve Gastrectomy (Experimental)
  Interventions: Procedure: Hand-Sewn Sleeve Gastrectomy
- Stapled Sleeve Gastrectomy (Active Comparator)
  Interventions: Procedure: Stapled Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Hand-Sewn Sleeve Gastrectomy — After laparoscopic sleeve gastrectomy, gastrectomy site is hand-sewn with 3/0 polypropylene suture and the specimen is removed transorally.
  Arms: Hand-Sewn Sleeve Gastrectomy
Procedure: Stapled Sleeve Gastrectomy — Laparoscopic sleeve gastrectomy is performed via 60 mm linear stapler (Endo GIATM Ultra, Covidien) .
  Arms: Stapled Sleeve Gastrectomy

SUMMARY:
Sleeve gastrectomy is a stapler dependent bariatric procedure. A hand-sewn sleeve gastrectomy can be necessary under certain circumstances. Here, the investigatorsaimed to compare the outcomes of hand-sewn and stapled sleeve gastrectomies for the first time.

In the hand-sewn group, no staplers were used and after vertical resection of the stomach by energy devices, the remnant stomach was closed by two rows intracorporeal sutures. In the stapler group, sleeve gastrectomy was done in the usual way.

DETAILED DESCRIPTION:
Nowadays, morbid obesity is a major health problem that the investigatorsface in every age groups. In the treatment of morbid obesity, sleeve gastrectomy is applied more and more frequently. However, sleeve gastrectomy is a stapler dependent operation and sleeve gastrectomy without the use of staplers was very limited in the literature [1]. Hand-sewn sleeve gastrectomy can rarely be necessary in some special conditions such as technical defects of the staplers, patients allergies to titanium clips or sometimes when staplers were unusable [1]. As far as the investigatorsknow, there was no study that compare the results of stapled and hand-sewn sleeve gastrectomies so far. The purpose of this study was to compare the hand-sewn and stapled sleeve gastrectomies in a small case series.

In June 2013, the investigatorslaunched a natural orifice surgery program including several procedures. In this context, the investigatorsplanned natural orifice (transoral) extraction of sleeve gastrectomy specimens. Patients who were eligible and agree with participation to the hand-sewn sleeve gastectomy combine with transoral specimen extraction study were accepted to two group. This study is conducted according to the STROCSS criteria. Total six morbidly obese patients (body mass index more than 40 kg/m2) who had undergone hand-sewn sleeve gastrectomy between the dates May-2014 and December 2014, were investigated retrospectively. In the same time period, seven another morbidly obese patients included in the control group were treated with stapled sleeve gastrectomies. Grouping was done by the acceptance of the patients. The hand-sewn sleeve gastrectomy group combined with natural orifice surgery. Patients who do not participate the hand-sewn group were treated by the stapled sleeve gastrectomy and the specimens were extracted through the trocar site. In both groups, patients' age, gender, height, weight, body mass index, comorbidity, and lifestyle properties were recorded. Intraoperative blood loss, operating time, length of hospital stay, postoperative complications, and the metabolic/bariatric results of the two groups in one and three years were evaluated. Statistical comparisons were performed with nonparametric statistical tests (Mann-Whitney U-test and Wilcoxon Signed Rank Test to analyze numerical data, and Fisher exact test to analyze cathegorical data). Numerical data expressed as median and range. P<0.05 was considered as significant.

In the hand-sewn group, following pneumoperitoneum with a Veres needle, the first 5 mm trocar was entered 14 cm down and 4 cm left from the xyphoid process. Other two 5 mm trocars were applied to the left and right upper quadrant. Last two 5 mm trocars were placed just below the xyphoid process for automatic liver retractor and through the epigastrium as a working port. A 5 mm 300 optic camera was used and the intraabdominal pressure was set to 14 mmHg. Gastrocolic and gastrosplenic ligaments were divided by 5 mm Ligasure (Force Triad, Covidien, Boulder, CO, USA) starting from 4-6 cm to pylorus till the angle of His. The greater curvature was liberated up to the left crus of the diaphragm. The anterior and posterior wall of the stomach were transected with a 5 mm Ligasure device under the guidance of a 36 F bougie, starting 4-6 cm away from the pylorus and division of both gatric leaves headed vertically in the direction of angle of His. After completion of the gastric division, the resected specimen was removed through the mouth with the help of an intraoperative peroral endoscopy using an endoscopic snare. The remaining open anterior and posterior walls of the stomach was continiously sutured each other by 3/0 polypropylene sutures. The suture length was 20 cm.

All the trocars were 5 mm in size in the hand-sewn group. The surgical technique of the stapled group has been defined in detail before (2). In short, vertical gastrectomy was applied with a 60 mm. lineer stapler (Endo GIATM Ultra, Covidien) under the guidance of 36 F bougie. These procedures were done through three 12 mm and two 5 mm trocars, that were placed to the same locations with the hand-sewn group. The specimen in the stapler group were extracted from the left upper quadrant trocar site. No supportive material or suture was use to the staple lines. Methylene blue test was done and a drain was place in all case.

After 6-8 hours postoperatively, the patients were mobilized, thromboembolic stockings were kept for five days. A liquid diet was started on day one. Prophylaxis of deep vein thrombosis was continued for 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of morbid obesity (body mass index over 40 kg/m2)
* Bariatric surgery must be the final decision of the obesity council.

Exclusion Criteria:

* Patients under legal age (<18 years)

Ages: 21 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-05-01; Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Volume of intraoperative blood loss | Depending on duration of the operation (60-300 mins)
  Intraoperative blood loss depending on duration of the operation (10-190 cc)
Duration of the operation | Depending on the type of the operation (60-300 mins)
  Operating time is compared between hand-sewn and stapled group

SECONDARY OUTCOMES:
Length of hospital stay | 3-10 days
  Postoperative length of hospital stay
Presence of postoperative complications | 3-13 days after the operation
  leakage, peritonitis, gastrointestinal haemorrhage

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT03982823/Prot_SAP_000.pdf